CLINICAL TRIAL: NCT00419978
Title: The Significance of Sentinel Node Analysis in Colon Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrural to study.
Sponsor: Legacy Health System (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 750040399
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colectomy

INTERVENTIONS:
Procedure: Colectomy

SUMMARY:
This study is for the patient with colon cancer, who is going to have colon cancer surgery. The purpose of this research study is to examine a specific lymph node, called the sentinel node. Lymph nodes are located throughout your body and cancer may spread by means of those lymph nodes. The sentinel node is the one located closest to your tumor. This study will find out if examining the sentinel node can help to predict disease progression. Since the value of this exam is unknown, taking part in this study will not change your clinical care.

ELIGIBILITY:
Inclusion Criteria:

* All patients must consent to participate in study
* Patients will be tracked for five years
* A blood test (CEA) will be collected every six months
* A CT scan will be performed annually
* A colonoscopy will be performed at 1 and 5 years post-surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-06; Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Whiteford, MD, Principal Investigator — Legayc Health System
Locations (1):
- Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon, United States

REFERENCES:
- See also: Legacy's internet website — http://www.legacyhealth.org